CLINICAL TRIAL: NCT02810327
Title: Alpha-1 Carrier Genomics Study
Status: Completed | Type: Observational
Sponsor: Medical University of South Carolina (Other)
Collaborators: CSL Behring (Industry)
Responsible Party: Sponsor
Other Study IDs: Pro00036911
Record Dates: First submitted 2016-06-20; First posted 2016-06-22 (Estimated); Results first posted 2019-07-22 (Actual); Last update posted 2019-07-22 (Actual); Status verified 2019-05

CONDITIONS: Alpha-1 Antitrypsin Deficiency; Emphysema; COPD; Smoking
Keywords: Alpha-1 antitrypsin deficiency; AATD; Alpha-1; SERPINA1; MZ; Carrier; Heterozygote; Smoking; COPD; Emphysema; Sequencing
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency; Emphysema; Pulmonary Disease, Chronic Obstructive; Smoking

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Bloodspot collections for DNA and limited protein analysis
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- MZ heterozygote with symptoms of COPD: Individuals who have previously had testing for Alpha-1 antitrypsin deficiency with genotype MZ (PiMZ) results. Individuals in this cohort have symptoms or clinical diagnosis of COPD.
  Interventions: Genetic: Genetic Sequencing
- MZ heterozygote without symptoms of COPD: Individuals who have previously had testing for Alpha-1 antitrypsin deficiency with genotype MZ (PiMZ) results. Individuals in this cohort do not have symptoms or clinical diagnosis of COPD.
  Interventions: Genetic: Genetic Sequencing

INTERVENTIONS:
Genetic: Genetic Sequencing — Sequencing of the SERPINA1 gene

SUMMARY:
The goal of this study is to better understand why some Alpha-1 genotype MZ (PiMZ) individuals develop chronic obstructive pulmonary disease (COPD) while others do not. This study will examine portions of the Alpha-1 gene that are not routinely tested to determine whether other changes in this gene correlate with development and progression of COPD. Participation involves responding to questionnaires about lung health and history, and performing an at-home finger stick to obtain blood spots using a test kit that is mailed. The blood provided will be used for genetic testing and correlation of results with COPD history. Participants will receive their results and access to genetic counseling at the conclusion of the study.

DETAILED DESCRIPTION:
Alpha-1 Antitrypsin Deficiency (AATD, Alpha-1) is the best established genetic risk factor for chronic obstructive pulmonary disease (COPD) and liver disease. Clinical presentation is heterogeneous in most genotypic populations of alpha-1 antitrypsin deficiency (AATD) and genetic variation in the Alpha-1 gene has been incompletely studied. Rare gene alterations that predispose to COPD risks of classic AATD in individuals without a classic homozygous deficiency genotype have not been studied and are important in understanding, testing and treating at-risk populations. Investigators hypothesize that SERPINA1 gene sequencing will find important sequence variations in previously assessed MZ individuals who have COPD compared to age, race, sex, AAT level and smoking status matched MZ individuals who do not have COPD.

The Alpha-1 Carrier Genomics study is a pilot study that will enroll up to 150 MZ individuals. COPD+ and COPD- individuals will be matched on age, sex, race and smoking history. Presence and severity of COPD is assessed by a COPD severity score on questionnaires. Participants will be mailed a test kit to obtain and return a blood sample by finger stick for the purpose of SERPINA1 gene sequencing. Gene sequencing will identify, if present, genomic signatures that may correlate with COPD in this cohort. Participants will receive their results and access to genetic counseling at the conclusion of this study.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. PiMZ individuals who fall into the lower quartile of AAT levels.

Exclusion Criteria:

1. Age <18 years
2. Known homozygous or compound heterozygous classic severe AATD (e.g. PiSZ, ZZ, Znull)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals age 18 and over who have previously had testing for Alpha-1 antitrypsin deficiency with genotype MZ (PiMZ) results, and an alpha-1 antitrypsin level of less than 16.0uM (83mg/dL) are eligible to participate.
Sampling Method: Non-Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charlie Strange, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina. Division of Pulmonary and Critical Care Medicine, Charleston, South Carolina, United States

REFERENCES:
- [Background] Demeo DL, Sandhaus RA, Barker AF, Brantly ML, Eden E, McElvaney NG, Rennard S, Burchard E, Stocks JM, Stoller JK, Strange C, Turino GM, Campbell EJ, Silverman EK. Determinants of airflow obstruction in severe alpha-1-antitrypsin deficiency. Thorax. 2007 Sep;62(9):806-13. doi: 10.1136/thx.2006.075846. Epub 2007 Mar 27. PMID 17389752
- [Background] Molloy K, Hersh CP, Morris VB, Carroll TP, O'Connor CA, Lasky-Su JA, Greene CM, O'Neill SJ, Silverman EK, McElvaney NG. Clarification of the risk of chronic obstructive pulmonary disease in alpha1-antitrypsin deficiency PiMZ heterozygotes. Am J Respir Crit Care Med. 2014 Feb 15;189(4):419-27. doi: 10.1164/rccm.201311-1984OC. PMID 24428606
- [Background] Eisner MD, Trupin L, Katz PP, Yelin EH, Earnest G, Balmes J, Blanc PD. Development and validation of a survey-based COPD severity score. Chest. 2005 Jun;127(6):1890-7. doi: 10.1378/chest.127.6.1890. PMID 15947299
- [Derived] Foil KE, Blanton MG, Sanders C, Kim J, Al Ashry HS, Kumbhare S, Strange C. Sequencing Alpha-1 MZ Individuals Shows Frequent Biallelic Mutations. Pulm Med. 2018 Sep 5;2018:2836389. doi: 10.1155/2018/2836389. eCollection 2018. PMID 30254761

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MZ Heterozygote With Symptoms of COPD | MZ Heterozygote Without Symptoms of COPD
Started | 76 | 41
Completed | 69 | 34
Not Completed | 7 | 7

BASELINE CHARACTERISTICS:
Population: Individuals age 18 and over with previous MZ results for Alpha-1 antitrypsin deficiency and AAT level in the lower MZ quartile (<16uM).
Groups:
- Total: Total of all reporting groups
Arm/Group | MZ Heterozygote With Symptoms of COPD | MZ Heterozygote Without Symptoms of COPD | Total
Number analyzed (Participants) | 76 | 41 | 117
Age, Continuous [Mean (Full Range); unit: years] — Population: 14 consented participants did not return their test kits and/or questionnaires.
  years
    Age: number analyzed (Participants) | 69 | 34 | 103
    Age | 51.7 [18 to 73] | 52.8 [29 to 70] | 52 [18 to 73]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 14 consented participants did not return their test kits and/or questionnaires.
  Participants
    number analyzed (Participants) | 69 | 34 | 103
    Female | 50 | 28 | 78
    Male | 19 | 6 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: 14 consented participants did not return their test kits and/or questionnaires.
  Participants
    number analyzed (Participants) | 69 | 34 | 103
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 1 | 0 | 1
    White | 68 | 34 | 102
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Abnormal Sequences in SERPINA1 Genes
Description: Additional SERPINA1 variant of known or possible significance detected by next generation sequencing.
Time Frame: End of study NGS Result
Measure: Number; unit: participants
Units Other Than Participants: samples
Arm/Group | MZ Heterozygote With Symptoms of COPD | MZ Heterozygote Without Symptoms of COPD
Number analyzed (Participants) | 69 | 34
Number analyzed (samples) | 69 | 34
participants | 6 | 0
Statistical Analysis 1: Comparison: MZ Heterozygote With Symptoms of COPD vs MZ Heterozygote Without Symptoms of COPD; The MUSC Bioinformatics Core analyzed group genomic data for variant association with COPD severity score, including single variant association or type of variant association with symptoms. Descriptive statistical analysis was performed using statistical package SAS 9.4 for Windows (SAS Institute Inc., Cary, NC, USA); Test type: Other; p = 0.054, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 1 year, 1 month
Arm/Group | MZ Heterozygote With Symptoms of COPD | MZ Heterozygote Without Symptoms of COPD
All-Cause Mortality (participants affected / at risk) | 0/76 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/76 | 0/41
Other Adverse Events (participants affected / at risk) | 0/76 | 0/41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2016-04-01): https://cdn.clinicaltrials.gov/large-docs/27/NCT02810327/Prot_000.pdf
  • Informed Consent Form (2016-05-12): https://cdn.clinicaltrials.gov/large-docs/27/NCT02810327/ICF_001.pdf
  • Statistical Analysis Plan (2016-04-01): https://cdn.clinicaltrials.gov/large-docs/27/NCT02810327/SAP_002.pdf